CLINICAL TRIAL: NCT07038434
Title: Refining mUltiple Artificial intelliGence strateGies for Automatic Pain Assessment Investigations: RUGGI Study
Acronym: RUGGI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valentina Cerrone (Other)
Collaborators: University of Salerno, Italy (Unknown); Federico II University (Other)
Responsible Party: Sponsor-Investigator, Valentina Cerrone, Study Coordinator, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Organization: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOURUGGI-0012506-2025
Record Dates: First submitted 2025-05-19; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Cancer Pain; Neuropathic Pain; Pain Assessment
Keywords: Artificial Intelligence; Machine Learning; Deep Learning; Automatic Pain Assessment; Facial Expression Analysis; Natural Language Processing; Stroop Test; Bio-signals; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Cancer Pain; Neuralgia

STUDY DESIGN:
Intervention Model Description: All participants receive the same diagnostic evaluation protocol, including clinical pain assessment, wearable bio-signal monitoring, neurocognitive testing, facial expression analysis, and language processing. The study is designed as a single-arm exploratory diagnostic protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-Based Pain Assessment in Chronic Pain Patients (Experimental): Participants with chronic pain will undergo a multimodal, non-invasive diagnostic assessment including self-reported pain questionnaires (NRS, DN-4, BPI), wearable biosignal acquisition (EEG, EMG, EDA, HRV), facial thermography using the HIRA system, video-based facial expression analysis, linguistic evaluation, and the Stroop Test. These data will be used to develop and validate machine learning models for automatic pain assessment.
  Interventions: Diagnostic Test: Multimodal AI-Based Pain Assessment

INTERVENTIONS:
Diagnostic Test: Multimodal AI-Based Pain Assessment — A non-invasive, multimodal diagnostic procedure combining self-reported pain scales (NRS, DN-4, BPI), wearable biosignal acquisition (EDA, EMG, HRV, EEG), facial thermography (HIRA system), video-based facial expression analysis, linguistic interview, and the Stroop Test. Data are used to train and validate machine learning models for automatic pain assessment in chronic pain patients.
  Other Names: Automatic Pain Assessment; AI Pain Evaluation

SUMMARY:
This single-center, non-profit, observational-interventional study aims to develop artificial intelligence (AI) models for the automatic assessment of chronic pain (APA - Automatic Pain Assessment). The study will enroll adult patients with chronic pain of various origins (oncologic and non-oncologic). Participants will undergo multidimensional evaluations that include clinical assessments, self-report questionnaires, bio-signal collection (e.g., EEG, EDA, HRV, GSR, PPG), and facial expression analysis via infrared thermography and video recordings.

The primary objective is to calibrate and test machine learning and deep learning models to recognize and predict the presence and severity of pain using multimodal data inputs. Secondary objectives include evaluating the effectiveness of pain treatments, assessing quality of life, and developing a standardized APA dataset for future research.

All data collection procedures are non-invasive and safe, and include tools like wearable sensors and standardized neurocognitive tests. The study is approved by the Italian Ethics Committee (Comitato Etico Territoriale Campania 2) and complies with GDPR and EU AI regulations.

DETAILED DESCRIPTION:
This study, titled "Refining mUltiple artificial intelliGence strateGies for automatic pain assessment Investigations" (RUGGI), explores the integration of AI in chronic pain evaluation. Pain is a multidimensional and subjective experience, and conventional assessment methods often rely solely on self-reported scales. This introduces the risk of over- or under-treatment. To overcome this limitation, the study leverages multimodal data-including physiological signals, facial expressions, and linguistic analysis-to build models capable of objectively assessing pain intensity and characteristics.

The primary aim is to calibrate predictive models (e.g., Support Vector Machines, Random Forest, Convolutional Neural Networks, YOLO architectures, and MLPs) that can recognize pain patterns using supervised and unsupervised learning. Bio-signals (EEG, HRV, GSR, EMG), infrared thermography (HIRA system), and prosodic-linguistic features will be analyzed. Data will be collected during structured timepoints: baseline (rest), Stroop test execution, and follow-up.

Patients are recruited based on chronic pain diagnosis per IASP and ICD-11 criteria. Inclusion criteria include age ≥18 and informed consent. The study foresees a target enrollment of approximately 200 patients within 6 months. Data will be processed following a rigorous AI pipeline, including preprocessing, feature extraction, dimensionality reduction, and cross-validation (k-fold with grid search optimization). Outcome measures include the Area Under the Curve (AUC), sensitivity, specificity, F1 score, and model explainability (via SHAP, LIME).

Secondary outcomes include assessing patient-reported quality of life, evaluating analgesic strategies, and generating a public-use APA dataset. All procedures are compliant with Good Clinical Practice (GCP), GDPR, and EU Artificial Intelligence Act (Reg. 2024/1689). The study is conducted at the University Hospital "San Giovanni di Dio e Ruggi d'Aragona" in Salerno, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with chronic pain, defined according to IASP and ICD-11 as pain that persists or recurs for more than three months.
* Diagnosed with either:
* Chronic primary pain (e.g., fibromyalgia, irritable bowel syndrome, chronic headaches)
* Chronic secondary non-cancer pain (e.g., low back pain, osteoarthritis, post-surgical pain)
* Chronic cancer-related pain (due to cancer or its treatment)
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Current treatment with psychotropic drugs or presence of active psychiatric disorders (e.g., psychosis, major depression).
* Known history of alcohol or substance abuse.
* Pregnancy or breastfeeding.
* Age under 18 years.
* Inability to provide informed consent (e.g., due to cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI models in classifying chronic pain | From Day 0 (baseline) to Day 30 (follow-up)
  Accuracy will be calculated to evaluate how well supervised machine learning and deep learning models can correctly classify the presence of chronic pain using multimodal data (e.g., biosignals, facial thermography, video, and audio).
Sensitivity of AI models in classifying chronic pain | From Day 0 to Day 30
  Sensitivity (true positive rate) will be computed to determine the model's ability to correctly identify patients experiencing chronic pain.
  Unit of measure: Sensitivity (%)
Specificity of AI models in classifying chronic pain | From Day 0 to Day 30
  Specificity (true negative rate) will be computed to assess the model's ability to correctly identify patients who are not experiencing chronic pain.
  Unit of measure: Specificity (%)
Precision of AI models in classifying chronic pain | From Day 0 to Day 30
  Precision (positive predictive value) will be calculated to assess the proportion of correct positive predictions among all positive classifications.
  Unit of measure: Precision (%)
F1-score of AI models in classifying chronic pain | From Day 0 to Day 30
  F1-score, the harmonic mean of precision and sensitivity, will be used to assess overall model performance, especially in the presence of class imbalance.
  Unit of measure: F1-score (numeric value)
AUC-ROC of AI models in classifying chronic pain | From Day 0 to Day 30
  The area under the receiver operating characteristic curve (AUC-ROC) will be used to evaluate the model's ability to discriminate between pain and no-pain conditions across thresholds.
  Unit of measure: AUC-ROC (numeric value from 0 to 1)

SECONDARY OUTCOMES:
Change in Patient Global Impression of Change (PGIC) score | From Day 0 to Day 30
  This outcome will measure patients' perceived improvement in their condition using the PGIC scale.
  Unit of measure: Score on a 7-point Likert scale (1 = No change to 7 = Very much improved)
Change in Brief Pain Inventory (BPI) interference score | From Day 0 to Day 30
  This outcome will measure how much pain interferes with daily functioning, using the BPI interference subscale.
  Unit of measure: Score from 0 (no interference) to 10 (complete interference)
Correlation between analgesic treatments and pain intensity (NRS) | From Day 0 to Day 30
  The outcome will assess the correlation between the type and frequency of analgesic treatments and changes in pain intensity, measured with the Numeric Rating Scale (NRS).
  Unit of measure: Pearson correlation coefficient (r), NRS scores from 0 to 10

OTHER OUTCOMES:
Creation of a structured multimodal dataset for AI-based pain research | From Day 0 to Day 30
  A standardized and anonymized dataset will be developed from collected multimodal inputs (biosignals, thermography, facial videos, linguistic data, questionnaires) to enable future research.
  Unit of measure: Dataset availability (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cascella, MD, PhD, Principal Investigator — University of Salerno
Locations (1):
- Azienda Ospedaliera Universitaria San Giovanni di Dio e Ruggi d'Aragona, Salerno, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of biometric and video-derived data, including facial thermography and audio recordings. Although all data are anonymized, there remains a potential risk of re-identification through multimodal signals. Additionally, no specific provisions for data sharing were included in the original informed consent approved by the ethics committee.

REFERENCES:
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Cascella M, Di Gennaro P, Crispo A, Vittori A, Petrucci E, Sciorio F, Marinangeli F, Ponsiglione AM, Romano M, Ovetta C, Ottaiano A, Sabbatino F, Perri F, Piazza O, Coluccia S. Advancing the integration of biosignal-based automated pain assessment methods into a comprehensive model for addressing cancer pain. BMC Palliat Care. 2024 Aug 3;23(1):198. doi: 10.1186/s12904-024-01526-z. PMID 39097739
- [Background] Machova K, Szaboova M, Paralic J, Micko J. Detection of emotion by text analysis using machine learning. Front Psychol. 2023 Sep 20;14:1190326. doi: 10.3389/fpsyg.2023.1190326. eCollection 2023. PMID 37799520
- [Background] Albashayreh A, Bandyopadhyay A, Zeinali N, Zhang M, Fan W, Gilbertson White S. Natural Language Processing Accurately Differentiates Cancer Symptom Information in Electronic Health Record Narratives. JCO Clin Cancer Inform. 2024 Aug;8:e2300235. doi: 10.1200/CCI.23.00235. PMID 39116379
- [Background] Lotsch J, Ultsch A, Mayer B, Kringel D. Artificial intelligence and machine learning in pain research: a data scientometric analysis. Pain Rep. 2022 Nov 3;7(6):e1044. doi: 10.1097/PR9.0000000000001044. eCollection 2022 Nov-Dec. PMID 36348668
- [Background] Cascella M, Schiavo D, Cuomo A, Ottaiano A, Perri F, Patrone R, Migliarelli S, Bignami EG, Vittori A, Cutugno F. Artificial Intelligence for Automatic Pain Assessment: Research Methods and Perspectives. Pain Res Manag. 2023 Jun 28;2023:6018736. doi: 10.1155/2023/6018736. eCollection 2023. PMID 37416623
- [Background] Nicholas MK. The biopsychosocial model of pain 40 years on: time for a reappraisal? Pain. 2022 Nov 1;163(Suppl 1):S3-S14. doi: 10.1097/j.pain.0000000000002654. No abstract available. PMID 36252231
- [Background] Kutafina E, Becker S, Namer B. Measuring pain and nociception: Through the glasses of a computational scientist. Transdisciplinary overview of methods. Front Netw Physiol. 2023 Feb 10;3:1099282. doi: 10.3389/fnetp.2023.1099282. eCollection 2023. PMID 36926544
- [Background] Lang VA, Lundh T, Ortiz-Catalan M. Mathematical and Computational Models for Pain: A Systematic Review. Pain Med. 2021 Dec 11;22(12):2806-2817. doi: 10.1093/pm/pnab177. PMID 34051102
- [Background] Kaplan CM, Kelleher E, Irani A, Schrepf A, Clauw DJ, Harte SE. Deciphering nociplastic pain: clinical features, risk factors and potential mechanisms. Nat Rev Neurol. 2024 Jun;20(6):347-363. doi: 10.1038/s41582-024-00966-8. Epub 2024 May 16. PMID 38755449
- [Background] Clauw DJ. From fibrositis to fibromyalgia to nociplastic pain: how rheumatology helped get us here and where do we go from here? Ann Rheum Dis. 2024 Oct 21;83(11):1421-1427. doi: 10.1136/ard-2023-225327. PMID 39107083
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Rahman S, Kidwai A, Rakhamimova E, Elias M, Caldwell W, Bergese SD. Clinical Diagnosis and Treatment of Chronic Pain. Diagnostics (Basel). 2023 Dec 18;13(24):3689. doi: 10.3390/diagnostics13243689. PMID 38132273
- [Background] Zimmer Z, Fraser K, Grol-Prokopczyk H, Zajacova A. A global study of pain prevalence across 52 countries: examining the role of country-level contextual factors. Pain. 2022 Sep 1;163(9):1740-1750. doi: 10.1097/j.pain.0000000000002557. Epub 2021 Dec 15. PMID 35027516